CLINICAL TRIAL: NCT05201508
Title: Sutures Only Versus Absorbable Polyglactin (Vicryl®) Mesh in Closure of Hiatal Defect in Laparoscopic Paraesophageal Hernia Repair: Randomized Controlled Trial.
Brief Title: Sutures Versus Polyglactin Mesh in Hiatal Hernia Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Collaborators: Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Olli Helminen, MD, PhD, Adjunct professor, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sutures or mesh for PEH
Record Dates: First submitted 2021-12-16; First posted 2022-01-21 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Paraesophageal Hernia; Hiatal Hernia; Hiatal Hernia, Paraesophageal; Recurrence
MeSH Terms: conditions — Hernia, Hiatal; Recurrence

STUDY DESIGN:
Intervention Model Description: Prospective open label randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sutures only (Active Comparator): Traditional suture closure of hiatal defect
  Interventions: Procedure: Sutures only
- Polyglactin mesh (Experimental): In addition to traditional sutures, key hole polyglactin mesh for hiatal defect closure.
  Interventions: Procedure: Polyglactin mesh

INTERVENTIONS:
Procedure: Polyglactin mesh — Polyglactin mesh is used in keyhole manner to enforce hiatal closure
  Arms: Polyglactin mesh
Procedure: Sutures only — Traditional hiatal closure with non-absorbable sutures.
  Arms: Sutures only

SUMMARY:
Paraesophageal hernia causes pain, heartburn, regurgitation, anemia and in extreme, life-threatening strangulation. For symptomatic patients, laparoscopic surgery is offered which includes hiatal defect closure and antireflux surgery. However, recurrence rates are high between 12 and 42%. In order to reduce recurrences, mesh has been used with various materials and techniques with conflicting results. Non-absorbable mesh has been linked with adverse events including erosion of esophageal wall. Traditionally used biological mesh materials are expensive and therefore problematic in routine use. Use of polyglactin (Vicryl®) mesh, which degrades in 6-8 week, has been reported in paraesophageal hernia surgery. Previously, no randomized controlled trial comparing sutures only and polyglactin mesh has been performed. In this trial, the aim was to randomize total of 110 patients to receive sutures only or mesh repair. Primary outcome was recurrence of paraesophageal hernia at 6 months after the repair based on computed tomography scan. Secondary outcomes included symptomatic recurrences, reoperation rate, quality of life, reoperations up to 20-years after surgery and use of proton pump inhibitors up to 20-years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Type III-IV PEH with either radiologic or endoscopic confirmation
* Scheduled for laparoscopic PEH repair
* The informed consent is acquired

Exclusion Criteria:

* Need for esophagus lengthening procedure (Collis gastroplasty)
* Recurrent PEH
* Emergency surgery
* No written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2043-01-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic recurrence of PEH | 6 months after surgery
  Computed tomography based recurrence after sutures only versus polyglactin mesh

SECONDARY OUTCOMES:
Symptomatic versus asymptomatic recurrence rates | 6 months
  Symptomatic versus asymptomatic recurrence rates based on symptoms and radiographic finding
Reoperation rate | 20 years
  Reoperation rate related to hiatal hernia recurrence
Health related quality of life based on score in esophago-gastric questionnaire (EORTC qlq-og25) | 6 months
  The impact of PEH repair method to health-related quality of life score in esophago-gastric questionnaire (EORTC qlq-og25) at 6 months compared to preoperative level. Score is given between 25 and 100 points with higher score meaning worse quality of life.
Hiatal defect size related to recurrence rate | 6 months
  The correlation with size of hiatal defect (cm^2) to recurrence rate (scatter plot with defect size in x-axis and recurrent hernias in y-axis)
BMI and the risk of recurrence | 6 months
  The correlation of BMI to recurrence rate (scatter plot with BMI in x-axis and recurrent hernias in y-axis)
Proton pump inhibitor (PPI) use | 20 years
  Use on proton pump inhibitors at 1- 3-, 5-, 10- and 20-years after surgery related to intervention method (sutures only or polyglactin mesh)
Age and the risk of recurrence | 6 months
  The correlation of age (years) to recurrence rate (scatter plot with age in x-axis and recurrent hernias in y-axis)
Albumin level and the risk of recurrence | 6 months
  The correlation of nutritional status (albumin level) to recurrence rate (scatter plot with albumin in x-axis and recurrent hernias in y-axis)

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No